CLINICAL TRIAL: NCT05842616
Title: Norepinephrine Titration In Patients With Sepsis Induced Encephalopathy: Cerebral Pulsatility Index Compared To Mean Arterial Blood Pressure Guided Protocol
Brief Title: Cerebral Pulsatility Index Compared To Mean Arterial Blood Pressure Guided Protocol In Sepsis Induced Encephalopathy:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Salah Salem, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35559/6/22
Record Dates: First submitted 2023-04-15; First posted 2023-05-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Sepsis; Norepinephrine; Encephalopathy
MeSH Terms: conditions — Sepsis; Brain Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial doppler pulsatility index guided protocol (Experimental): Norepinephrine titration that will be guided by Transcranial doppler (TCD) pulsatility index.
  Interventions: Other: Transcranial doppler pulsatility index guided protocol
- Mean arterial blood pressure guided protocol (Active Comparator): Norepinephrine titration that will be guided by Mean arterial blood pressure (MAP).
  Interventions: Other: Mean arterial blood pressure guided protocol

INTERVENTIONS:
Other: Transcranial doppler pulsatility index guided protocol — Norepinephrine titration that will be guided by Transcranial doppler pulsatility index.
  Arms: Transcranial doppler pulsatility index guided protocol
Other: Mean arterial blood pressure guided protocol — Norepinephrine titration that will be guided by Mean arterial blood pressure (MAP).
  Arms: Mean arterial blood pressure guided protocol

SUMMARY:
The aim of our study is to compare between transcranial doppler pulsatility index and mean arterial blood pressure in guiding management of sepsis induced encephalopathy.

DETAILED DESCRIPTION:
Sepsis induced encephalopathy is the most frequent sepsis related organ dysfunction. It appears early during the course of infection, often before any other organ involvement in up to 70% of hospitalized septic patients and is associated with significant change of cerebral circulation caused by redistribution of blood flow during sepsis that accompanies the abnormal inflammatory response during an infection, in absence of direct central nervous system involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Must had clinical diagnosis of sepsis induced encephalopathy.

Exclusion Criteria:

* Refusal to participate in the study.
* Cerebral infection.
* Known cerebral lesions (Neoplasm, Traumatic brain injury, Stroke, Ischemic or hemorrhagic cerebrovascular lesions, high intracranial pressure).
* Known severe carotid stenosis (>70％).
* Intoxication due to drugs.
* Pregnancy.
* Patients supported by intra-aortic balloon pumb (IABP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Intensive care unit (ICU) mortality | 28 day or till death which earlier
  Incidence of Intensive care unit (ICU) stay will be recorded

SECONDARY OUTCOMES:
Mean arterial pressure | 24 hours
  Fluid resuscitation will be started using crystalloids at a rate of 4 to 6 ml/kg with reevaluation after 15 minutes.
  If MAP is still less than 65 mmhg, fluid resuscitation should be continued at a rate of 4 to 6 ml/kg with reevaluation after another 15 minutes up to 30 ml/kg.
  Vasopressors will be started if the patient is still hypotensive during or after resuscitation without delay even peripherally to avoid delay until central venous access is secured (norepinephrine is the first line agent preferred over other vasopressors).
Norepinephrine titration | 24 hours
  Fluid resuscitation will be started using crystalloids at a rate of 4 to 6 ml/kg with reevaluation after 15 minutes.
  If MAP is still less than 65 mmhg, fluid resuscitation should be continued at a rate of 4 to 6 ml/kg with reevaluation after another 15 minutes up to 30 ml/kg.
  Vasopressors will be started if the patient is still hypotensive during or after resuscitation without delay even peripherally to avoid delay until central venous access is secured (norepinephrine is the first line agent preferred over other vasopressors).
Cerebral perfusion pressure | 24 hours
  Cerebral perfusion pressure (CPP) will be done using transcranial doppler.
Outcome of encephalopathy | 28 day
  Encephalopathy outcome at ICU discharge using Glasgow coma scale (GCS)
SOFA score | Up to 4 weeks.
  SOFA score at ICU admission and discharge.
Length of ICU stay | At least 28 days
  Length of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Mai S Aboshaara, MD, Principal Investigator — Assistant lecturer
Locations (1):
- Tanta University Hospitals, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol, SAP
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author

REFERENCES:
- [Derived] Salem MS, Abosabaa MA, Abd El Ghafar MS, Ei-Gendy HMEM, Alsherif SEI. Norepinephrine titration in patients with sepsis-induced encephalopathy: cerebral pulsatility index compared to mean arterial pressure guided protocol: randomized controlled trial. BMC Anesthesiol. 2025 Jan 4;25(1):5. doi: 10.1186/s12871-024-02814-0. PMID 39755598